CLINICAL TRIAL: NCT05598255
Title: Comparison of Caudal Blockade and Dorsal Penile Nerve Block With and Without the Intravenous Administration of Dexamethasone for Analgesia After Paediatric Male Circumcision: a Single Centre Randomized-controlled Trial
Brief Title: Comparison of Caudal Blockade and Dorsal Penile Nerve Block With and Without the Intravenous Administration of Dexamethasone for Analgesia After Paediatric Male Circumcision
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped early due to low recruitment, an extended projected timeline, and the need to transfer the study to CTIS, which made continuation unfeasible.
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Joris Goossens, MD, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MMS.2022.006
Record Dates: First submitted 2022-07-07; First posted 2022-10-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Analgesic Effect
Keywords: Locoregional technique; postoperative analgesic effects; caudal blockade; dorsal penile nerve block
MeSH Terms: interventions — Dexamethasone; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: patient and parents, recovery nurses and study nurse will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caudal blockade (with levobupivacaine) and dexamethasone IV (Active Comparator): Administration of levobupivacaine 0,25% 0,5 ml/kg through the hiatus sacralis lege artis. IV administration of dexamethasone 0,5mg/kg (max. 5mg) during standard anaesthetic management.
  Interventions: Drug: Dexamethasone; Procedure: Caudale Blockade with levobupivacaine
- Dorsal penile nerve block (with levobupivacaine) and dexamethasone IV (Active Comparator): Administration of levobupivacaine 0,5% 0,1ml/kg on each side of the midline as described in Hadzic's textbook of regional anaesthesia. IV administration of dexamethasone 0,5mg/kg (max. 5mg) during standard anaesthetic management.
  Interventions: Drug: Dexamethasone; Procedure: Dorsal penile nerve block with levobupivacaine
- Dorsal penile nerve block (with levobupivacaine) (Active Comparator): Administration of levobupivacaine 0,5% 0,1ml/kg on each side of the midline as described in Hadzic's textbook of regional anaesthesia.
  Interventions: Procedure: Dorsal penile nerve block with levobupivacaine

INTERVENTIONS:
Drug: Dexamethasone — During standard anaesthetic management: IV administration of dexamethasone (0,5mg/kg, with a maximum dose of 5mg).
  Arms: Caudal blockade (with levobupivacaine) and dexamethasone IV; Dorsal penile nerve block (with levobupivacaine) and dexamethasone IV
Procedure: Caudale Blockade with levobupivacaine — Administration of levobupivacaine 0,25%0,5ml/kg through the hiatus sacralis lege artis, before incision.
  Arms: Caudal blockade (with levobupivacaine) and dexamethasone IV
Procedure: Dorsal penile nerve block with levobupivacaine — Administration of levobupivacaine 0,5% 0,1ml/kg on each side of the midline as described in Hadzic's textbook of regional anaesthesia, before incision.
  Arms: Dorsal penile nerve block (with levobupivacaine); Dorsal penile nerve block (with levobupivacaine) and dexamethasone IV

SUMMARY:
Male infant circumcision is a frequently performed, but painful procedure. A variety of methods, both systemic and locoregional, have been developed to overcome postoperative pain after circumcision. It has been shown that local anesthetic techniques are more effective than opioids. Especially caudal block and dorsal penile nerve block provide adequate early analgesia (up to 2 hours) after circumcision.

Although the postoperative analgesic effects of CB and DPNB have been evaluated in literature before, these two techniques that are commonly used in circumcision surgery in the paediatric population, have not yet been compared when using DXM as an adjuvant in both methods. On the other hand, to our knowledge there is no evidence that indicates any other advantage than a reduced incidence in PONV when it comes to circumcision patients having a DNPB with IV DXM.

Therefore, this study aims to evaluate the analgesic effect of CB using levobupivacain with IV DXM compared to DPNB using levobupivacain with IV DXM and DPNB without IV DXM. It is questioned whether the addition of IV DXM to the DPNB might shift our standard of care towards a locoregional technique avoiding the neuraxial route, without losing the analgesic quality of the combination of a CB with IV DXM.

DETAILED DESCRIPTION:
All male infant patients, between ≥ 1 and < 7 years of age, undergoing circumcision will be randomized in a 1:1:1 ratio to the

1. Caudal blockade group with dexamethasone or;
2. Dorsal penile nerve block group with dexamethasone or;
3. Dorsal penile nerve block group withouth dexamethasone.

After induction of anaesthesia the allocated locoregional anaesthesia technique will be performed.

For the caudal blockade group levobupivacaine 0,25% 0,5ml/kg will be administered through the hiatus sacralis lege artis. After performing the caudal blocakde, IV administration of dexamethasone 0.5 mg/kg (max. 5 mg).

For the dorsal penile nerve block levobupivacaine 0,5% 0,1ml/kg will be administered on each side of the midline as described in Hadzic's textbook of regional anaesthesia. After performing of the dorsal penile nerve block, IV administration of dexamethasone 0.5 mg/kg (max. 5 mg) in patients in the dorsal penile nerve block group with dexamethasone .

IV administration of diclofenac 1mg/kg and paracetamol 15mg/kg for both groups. If heart rate raises with >20% from baseline within 2 minutes after incision, administration of sufentanyl (0,1µg/kg IV) is necessary.

Pain scores are evaluated after awakening at PACU, measured by the FLACC scale, at following timepoints: 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours and 24 hours postoperative. During recovery stay till hospital discharge pain scores will be registered by the study nurse. Registration of pain scores after hospital discharge (till 24 hours postoperative) will be performed by (one of) the parents of the patient, who will be educated how to use the FLACC scale by the study nurse. A follow up phone call will be performed by the study nurse to collect the remaining pain scores starting from hospital discharge.

Pain medication exists of standard administration of paracetamol PO 15mg/kg every 6 hours (starting 6 hours after the intraoperative administered dose) and ibuprofen PO 10mg/kg every 8 hours (starting 8 hours after the intraoperative administered diclofenac).

When FLACC score remains above 3, rescue pain medication will be administered during hospital stay. Rescue pain medication consists of tramadol intravenously (PACU) or oral drops (ward) 1mg/kg and can be repeated at maximum every 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male paediatric patients, between ≥ 1 and < 7 years of age
* Patients scheduled for paediatric male circumcision (sleeve resection technique)
* Signed written informed consent form

Exclusion Criteria:

* Patients known with allergy to study medication (in this case levobupivacaine, dexamethasone, tramadol, diclofenac, paracetamol, sufentanil)
* ASA score 3 or higher (ASA physical satus classification system)
* Delayed motor development/inability to stand up
* Patients who receive medication that could possibly interact with levobupivacaine (mexiletine, ketoconazole, theophylline)
* Patients who simultaneous participate in another interventional clinical trial
* Inability of parents to understand Dutch in a sufficient way
* Soft tissue infection in the area of the procedure
* Coagulation disorder
* Spina bifida
* Autism spectrum disorder
* Ulcus ventriculi and duodeni
* Systemic fungal, bacterial and parasitic infections
* Administration of live or live-attenuated vaccins during the use of dexamethasone

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic effect | 24 hours postoperative
  Analgesic effect of a caudal blockade after circumcision in paediatric patients compared to dorsal penile nerve block after circumcision in paediatric patients measured by the FLACC scale (= Face, Legs, Activity, Cry, Consolability) at 30 minutes, 1, 2, 6, 12 and 24 hours postoperative

SECONDARY OUTCOMES:
Need for escape analgesia | From PACU admission until hospital discharge (up to 48 hours)
  Need for escape analgesia, in this study tramadol
Incidence of nausea and vomiting (PONV) | From PACU admission until 24 hours postoperative
  Incidence of nausea and vomiting at 30 minutes, 1, 2, 6, 12 and 24 hours postoperative
Time to micturition | From PACU admission until hospital discharge (up to 48 hours) (measured every 30 minutes starting from PACU admission until hospital discharge)
  minutes
Total procedure time | perioperative
  minutes
Length of hospital stay | From hospital admission until hospital discharge (up to 48 hours)
  Hours
Time to standing up | From PACU admission until hospital discharge (up to 48 hours) (measured every 30 minutes starting from PACU admission until hospital discharge)
  minutes
Need for supplemental sufentanil intraoperatively | perioperative
  If heart rate raises with >20% from baseline within 2 minutes after incision, administration of sufentanil (0.1 µg/kg IV) is necessary

CONTACTS AND LOCATIONS:
Overall Officials: Joris Goossens, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares Gent, Ghent, Oost Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No